CLINICAL TRIAL: NCT05106166
Title: Joint Attention-Based Occupational Therapy Intervention in Pre-Schoolers With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Joint Attention-Based Occupational Therapy Intervention in Pre-Schoolers With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sümeyye Belhan Çelik, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/126
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder; Social Communication; Behavior Problem; Visual Perceptual Weakness
MeSH Terms: conditions — Autism Spectrum Disorder; Communication; Mental Disorders | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This prospective studies that measure the effectiveness of occupational therapy intervention. Randomized controlled trials (RCT) are prospective studies that measure the effectiveness of a new intervention or treatment. Participants are recruited and randomly assigned to either the intervention or the comparator group. It is important to ensure that at the time of recruitment there is no knowledge of which group the participant will be allocated to; this is known as concealment. It is examined whether there is any difference in the results of the study intervention and also the intervention and control group are compared.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: occupational therapy program + the usual special education program (USEP) (Experimental): The practitioner used the less-to-more orientation to get the child to respond to the offer of joint attention. For example, if the child did not respond to the joint attention offer within 5-10 seconds, practitioner first directed the child, used exaggerated gestures, gave a moving hint if he still did not respond, and physically slowly directed the child's head towards the target if he still did not respond. In addition, the practitioner gave a verbal command (practitioner said: look at how his arms are waving, pointing to the toy, now look at me). When the child looked at the toy and reacted, he again gave enthusiastic and activity-appropriate feedback (e.g. he tickled the child, saying, "Isn't it weird, is there ever such a long arm?"). The child's interest and leadership in the activities were followed, including what the child did and said. Positive feedback was then provided.
  Interventions: Behavioral: Occupational Therapy
- Control group: the usual special education program (USEP) (Active Comparator): The USEP studied was including gross motor skills, communication skills, preschool preparation skills, and self-care skills. The control group of the study consisted of children attending the USEP.
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Behavioral: Occupational Therapy — occupational therapy sessions are based on the joint attention

SUMMARY:
In order to support the development of preschool children, joint attention training with activities incorporated in their natural routines can support the achievement of occupational therapy goals. This study explores the adjunctive benefit of a joint attention-based occupational therapy program offered in addition to the usual special education program (USEP) compared to USEP alone.

The present study was designed as a randomized controlled study, including pre-post testing. The Social Communication Questionnaire (SCQ), Autism Behaviour Checklist (ABC), and A Motor-Free Visual Perception Test 4 (MVPT-4) were implemented to measure the participants' conditions before and after the intervention.

DETAILED DESCRIPTION:
Twenty children, ten in each group, were included in the study. The study inclusion criteria were being between the ages of 4 and 6, diagnosed with ASD, and consenting to participate in the study. The study did not include children who had a co-morbid condition other than ASD and had no previous education or training. Between 1 April and 25 June 2020, a total of 28 children were interviewed for this study, and 3 children were excluded because they did not meet the inclusion criteria. 13 children were randomly assigned to the study group and 12 children to the control group. 3 individuals from the study group were excluded because of time, transportation or other reasons, and 2 children from the control group were excluded because they did not complete the assessments. As a result, a total of 20 children with ASD, 10 of whom were working and 10 were control, formed the sample group of the study. Informed consent was obtained after the scope and purpose of the study were explained in detail to the participants and primary family caregivers.

A social communication questionnaire (SCQ), autistic behavior checklist (ABC), and motor-free visual perception test-4 (MVPT-4) were administered to the children before and after the intervention, and the results were compared.

The SCQ was developed to evaluate the social communication of individuals with autism. The total score can be between 0-and 39 for children who can speak. The SCQ which comprises three sub-dimensions: reciprocal social interaction, language and communication, and repetitive and stereotyped patterns has the validity and reliability in Turkish.

The ABC is among the scales used for screening and evaluating education in autism in many countries. The ABC consists of five sub-dimensions: sensory, relating, body or object use, language, and social and self-help. The total score is between 0-159.

MVPT-4 is an instrument that presents a fast, reliable, and valid evaluation of children and adults' general and visual perceptual abilities. MVPT-4 consists of 45 items that are organized and grouped to provide a smooth implementation process. The items consist of black and white drawings and patterns developed to present answer options, making the implementation easy in a multiple-choice form. Motor skills are not necessary to get a response, which makes this test useful, especially for people with motor disabilities.

All children included in the study attend a usual special education program (USEP) 2 sessions per week in a rehabilitation center. The USEP studied was including gross motor skills, communication skills, preschool preparation skills, and self-care skills. The control group of the study consisted of children attending the USEP. Children in the study group received an occupational therapy intervention based on joint attention in addition to the USEP they continued. As an intervention in the study group, the sessions were conducted three days a week for a total of 12 weeks. The initial assessments were administered to children in both groups. At the end of the 12 weeks, the evaluations were repeated in both groups.

The acquisition frame of reference, which proposes to shape the behaviors that contribute to skill acquisition, and the developmental frame of reference, which emphasizes the continuous change and emergence of skills with age, guided the occupational therapy intervention. Therefore, all activities were designed according to the chronological and developmental ages of the children. During the joint attention-based intervention sessions, holistic occupational therapy approaches for the child's sensory, physical, social, language and communication deficits were discussed.

The steps followed are:

1. Each parent was interviewed about the child's preferences. The toy types preferred by a child and the toys that a child might react negatively to were identified. The intervention specialist selected a total of 15 toys for paired stimulus preference assessments. Five of these toys were stuffed animals and figures. Five comprised multi-part activities, and the other five consisted of toys activated by light, movement, and/or sound. Each group of toys was used according to the child's interests and habits in three stages: creating a response to a joint attention offer, initiating joint attention, and reinforcing a joint attention response.
2. During the joint attention-based occupational therapy intervention, researchers paid attention to maintaining eye contact and following the child's lead. Activities were conducted at the desk and on the floor. A game pattern was created using the selected toys; the pattern was planned and implemented as activities for an average of 20 minutes.
3. In the sessions, (a) fine motor activities such as handicrafts, finger games; (b) gross motor activities such as obstacle course, music, dance; (c) visual-motor activities such as drawing, cutting, and assembly were used. Initiating and responding to joint attention during these activities was the focus of the intervention. With the training, the aim was to generalize behavioral skills and transfer them to the context of social play.
4. It is stated that compatible environmental arrangements that will provide visual cues are important when structuring environmental activities because children with autism respond to the use of visual input. For this reason, environmental arrangements were made with visual stimuli that could attract a child's attention.

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion criteria were being between the ages of 4 and 6
* diagnosed with ASD
* consenting to participate in the study.

Exclusion Criteria:

* The study did not include children who had a co-morbid condition other than ASD
* had no previous education or training.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Autistic Behavior Checklist (ABC) | 12 weeks
  The ABC is among the scales used for screening and evaluating education in autism in many countries. The ABC consists of five sub-dimensions: sensory, relating, body or object use, language, and social and self-help. The total score is between 0-159. Minimum score is 159. Maximum score is 0.

SECONDARY OUTCOMES:
Social Communication Questionnaire (SCQ) | 12 weeks
  The SCQ was developed to evaluate the social communication of individuals with autism. The total score can be between 0-and 39 for children who can speak. The SCQ which comprises three sub-dimensions: reciprocal social interaction, language and communication, and repetitive and stereotyped patterns. Minimum score is 39. Maximum score is 0.
Motor-free Visual Perception Test-4 (MVPT-4) | 12 weeks
  MVPT-4 is an instrument that presents a fast, reliable, and valid evaluation of children and adults' general and visual perceptual abilities. MVPT-4 consists of 45 items that are organized and grouped to provide a smooth implementation process. The items consist of black and white drawings and patterns developed to present answer options, making the implementation easy in a multiple-choice form. Motor skills are not necessary to get a response, which makes this test useful, especially for people with motor disabilities. Maximum score is 45. Minimum score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Belhan Çelik, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not planned to be shared to protect the privacy of the clients, but it can only be shared with the editor or the referee of the submitted journal if they want to see it.